CLINICAL TRIAL: NCT06802458
Title: The Effect of Motivational Interviewing on Healthy Lifestyle Behaviors and Quality of Life in on Menopausal Women: a Pilot Randomized Controlled Trial
Brief Title: Motivational Interviewing on Healthy Lifestyle Behaviors and Quality of Life in on Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: Munzur University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Head of Department of Women's Health and Disease Nursing, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03/09/2018/4579
Record Dates: First submitted 2025-01-17; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Menopause; Nursing
Keywords: motivational interviewing; healthy lifestyle behavior; menopause specific quality of life
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention)
- Experimental (Experimental)
  Interventions: Other: Motivational interviewing

INTERVENTIONS:
Other: Motivational interviewing — A total of 9 sessions were conducted, including 1 preparation session, 6 motivational interviews, 1 initial follow-up interview one week after the intervention, and 2 follow-up interviews 4 weeks after the initial follow-up. Considering the interactive training method, the motivational interviewing sessions were conducted in the training room of the Health Center in groups of 10 at three different days (Monday, Thursday, Friday) once a week, through face-to-face sessions each lasting 50-60 minutes. During the interviews, the women were provided with counseling to activate their own sources of motivation, develop healthy lifestyle behaviors and improve their quality of life specific to menopause
  Arms: Experimental

SUMMARY:
Background: This study aims to determine the effect of motivational interviewing on healthy lifestyle behaviors and quality of life in menopausal women.

Methods: This is a randomized controlled empirical study. The study was conducted with a total of 136 women, including 68 for experimental group and 68 for control group. The data were collected using an introductory information form, the Health Promoting Lifestyle Profile II (HPLPL II) and the Menopause-Specific Quality of Life (MENQOL). Women in the experimental group received 6 sessions of motivational interviewing and 2 follow-up interviews in two family health centers (FHCs) from the researcher. No intervention was applied to women in the control group. The data were analyzed using number, percentage, mean, standard deviation, chi-square test, Bonferroni test, independent samples t test and repeated ANOVA.

ELIGIBILITY:
Inclusion Criteria:

1. being literate;
2. being able to make a conscious decision to participate in the study, being able to communicate verbally, and being able to sign a consent form;
3. having had menopause naturally and within the last 3 years;
4. being sexually active;
5. having no hormone replacement therapy.

Exclusion Criteria:

1. unwilling to continue the study;
2. having a psychiatric diagnosis according to the FHC records.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Health Promoting Lifestyle Profile II | change from starting to 0. and 7. week
  The scale includes six dimensions, namely, nutrition, physical activity, stress management, interpersonal relationships, responsibility for health, and spiritual growth (52 items in total). The items are scored based on a 4 point Likert scale (never, sometimes, often, and usually). The total score of the scale ranges from 52 to 208. The score of each dimension is calculated separately and a higher scores mean better health.
Menopause-Specific Quality of Life | change from starting to 0. and 7. week
  This is a 7-point Likert-type scale containing 29 items and consists of four domains: vasomotor, psychosocial, physical and sexual. Each item is scored from "0" to "6", where "0" refers to "not bothersome" and "6" to "extremely bothersome". A higher scale score indicates greater severity of the complaint.

CONTACTS AND LOCATIONS:
Locations (1):
- Munzur University, Tunceli, Tunceli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Orhan I, Yagmur Y. The effect of motivational interviewing on healthy lifestyle behaviors and quality of life in on menopausal women: a pilot randomized controlled trial. BMC Womens Health. 2025 Jul 4;25(1):306. doi: 10.1186/s12905-025-03807-y. PMID 40611241